CLINICAL TRIAL: NCT03606850
Title: Pilot Study on the Identification of Cortical Excitability Changes Measured by Transcranial Magnetic Stimulation (TMS) as Markers of Antidepressant Response
Brief Title: Transcranial Magnetic Stimulation Study of Cortical Excitability as Marker of Antidepressant Response: EXCIPSY Study
Acronym: EXCIPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier du Rouvray (Other Government)
Collaborators: Centre hospitalier de Ville-Evrard, France (Other); University Hospital Caen, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00157-48
Record Dates: First submitted 2018-07-19; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Major Depressive Disorder
Keywords: cortical excitability; marker of response
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The patients will assess for markers of cortical excitability (cortical silent period CSP, resting motor threshold RMT, motor evoked potential MEP, intra-cortical inhibition ICI and intra-cortical facilitation ICF) before treatment, at day 3, day 7, day 14, day28 and day 60 with an assessment of depression (HAMD-21).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment by citalopram (Experimental): The patients will receive a treatment by citalopram at 20mg/day. If patients respond by at least 20% on the HAMD-21 scale at day 14 : continuation at 20 mg/day. If patients do not respond by at least 20% at day 14 : increase the dose at 40 mg/day. The patients who will not respond by at least 50% on the HAMD-21 scale at day 28 will be excluded of the study and will undergo a new treatment plan. The patients who will respond by at least 50% on HAMD-21 at day 28 will continue citalopram at the same dose and will be reappraised at day 60. The patients will be assessed for the markers of neuroexcitability at day 1, day 3, day 7, day 14, day 28 and day 60.
  Interventions: Device: Measurements of markers of cortical excitability by TMS

INTERVENTIONS:
Device: Measurements of markers of cortical excitability by TMS — In the arm experimental "treatment by citalopram", measurements of markers of cortical excitability by Transcranial Magnetic Stimulation will be applied. These measurements were: the cortical silent period CSP, the evoked potential MEP, the intra-cortical inhibition ICI and the intra-cortical facilitation ICF). Electromagnetic coil is placed upon the vertex, according to the International 10-20 EEG system. Gathering of the peripheral signal by a surface EMG electrode (non invasive device) placed regarding one of the first dorsal interosseous muscle.

SUMMARY:
Depression is a common issue but there is no marker of response to an antidepressant treatment.The measurement of variation of the cortical excitability in responders to a selective serotonin reuptake inhibitor (SSRI) (compared to no-responders) had never been done before. In the study of Robol et al. (2004) concerning the acute effects of citalopram on markers of cortical excitability, the authors have pointed out an increase on the cortical silent period (CSP) after administration of citalopram (2.5 hours). The investigators hypothesize that this effect remains later and that the diminution of cortical excitability could be a biomarker of antidepressant response. In this case, they expect that the variation of CSP between day 1 and day 28 is higher in responders to a SSRI (citalopram) compared to non-responders. the investigators lead a pilot, prospective, multicentric study in drug-naive patients to compare the variation of the markers of cortical excitability (the CSP but to the resting motor threshold RMT, the motor evoked potential MEP, the intra-cortical inhibition ICI and the intra-cortical facilitation ICF) between day 1 and day 28 in responders to citalopram, compared to non-responders.

ELIGIBILITY:
Inclusion criteria:

* major depressive episode (according to DSM 5 criteria). Severity of depressive episode assessed by Hamilton Depressive Rating Scale 21 items (HAMD-21) : score > 15 (significant impairment), low suicide risk (score < 2 on suicide item).
* Drug-naive patient (or antidepressant stopped for more than 3 months).
* Patient covered by security social system.
* Patient who is able to read and understand the information paper. Patient who is able to sign the consent.
* For women of childbearing age, effective method of contraception (estrogen-progestin contraceptive or intra-uterine device or tubal ligation) for more than 1 month (negative pregnancy test).

Exclusion criteria:

* Coprescription of psychoactive or neurological drugs known to alter cortical excitability
* Other psychiatric disorders (psychotic disorders, eating disorders).
* Change of antidepressive drug during the study.
* Abuse or addiction at other substances than nicotine or caffeine.
* Unsteady consumption of nicotine or caffeine.
* Dermatologic disease, dementia, medical history of seizure or epilepsy, brain tumor, metallic biomedical implants in brain.
* Ongoing treatment by magnetic or electric stimulation (for example : transcutaneous nerve stimulation or spinal cord stimulation).
* Women of childbearing age without effective contraception, pregnant or breastfeeding.
* Patient who was already included in a clinical trial within 30 days before the inclusion visit.
* Patient deprived of liberty and under guardianship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Variation of the CSP between day 1 and day 28 | 28 days
  The difference in variation of the cortical silent period (CSP) between day 1 and day 28 in responders compared to non-responders. A decrease by at least 50% on Hamilton Depression rating Scale (HAMD-21) define response to citalopram.The HAMD-21 assesses the intensity of the depressive symptoms with 21 items. Its score is between 0 (no depression) and 73 (the maximum of intensity).

SECONDARY OUTCOMES:
Variation of the RMT between day 1 and day 28 | 28 days
  The difference in variation of other markers of cortical excitability like resting motor threshold (RMT) between day 1 and day 28 in responders compared to non responders.
Variation of the MEP between day 1 and day 28 | 28 days
  The difference in variation of the motor evoked potential (MEP) between day 1 and day 28 in responders compared to non responders.
Variation of the ICI between day 1 and day 28 | 28 days
  The difference in variation of the intra-cortical inhibition (ICI) between day 1 and day 28 in responders compared to non responders.
Variation of the ICF between day 1 and day 28 | 28 days
  The difference in variation of the intra-cortical facilitation (ICF) between day 1 and day 28 in responders compared to non responders.
Variation of the markers of cortical excitability at other times | 14 days
  Differences in variations of RMT, MEP, ICI and ICF in responders compared to non-responders at other times : between day 1 and day 3, day 1 and day 7 and day 1 and day 14.
Variation in HAMD-21 between day 1 and day 60 for the responders at day 28 | 60 days
  The variation in HAMD-21 between day 1 and day 60 for the responders at day 28.
Variations in UKU (Udvalg pour Kliniske Undersøgelser Side Effect Rating Scale) at different times | 60 days
  The variations in UKU scale adapted for antidepressants at day 3, day 7, day 14, day 28 (and day 60 for the responders at day 28). The UKU assesses the side effects of the antidepressants. Its score is between 0 (no side effect) and 120 (the maximum of side effects).
Variations in Morisky compliance scale | 60 days
  The variations in Morisky compliance scale at day 3, day 7, day 14, day 28 (and day 60 for the responders at day 28).The Morisky scale assesses the compliance with antidepressant treatment and its score is between 0 (no compliance) and 8 (good compliance).

CONTACTS AND LOCATIONS:
Locations (1):
- Rouvray Hospital, Sotteville-lès-Rouen, France